CLINICAL TRIAL: NCT03687229
Title: The Effect Of Direct Acting Antiviral Drugs on miRNA-122 And Insulin Resistance In Chronic HCV Patients
Brief Title: The Effect Of DAAs on miRNA-122 And Insulin Resistance In Chronic HCV Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAAbdelmegid, Principal Investigastor, Assiut University
Other Study IDs: miRNA-122 in chronic HCV
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis c
Keywords: micro ribonucleic acid-122; insulin
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Chronic HCV patients before treatment & 3 months after starting of treatment. not known to be:
  1. Cirrhosis
  2. Diabetes Mellitus.
  3. Hemochromatosis
  4. HBV
  5. HIV.
  6. Hepatocellular carcinoma (HCC)
  7. Chemotherapy
  8. Organ transplantation
  Interventions: Diagnostic Test: A)microribonucleic acid-122(miRNA-122), B) Hepatitis C virus Real Time Polymerase chain Reaction (HCV RT-PCR); Diagnostic Test: A)fasting serum glucose, B)Fasting serum insulin
- Control: Apparently healthy individuals
  Interventions: Diagnostic Test: A)microribonucleic acid-122(miRNA-122), B) Hepatitis C virus Real Time Polymerase chain Reaction (HCV RT-PCR); Diagnostic Test: A)fasting serum glucose, B)Fasting serum insulin

INTERVENTIONS:
Diagnostic Test: A)microribonucleic acid-122(miRNA-122), B) Hepatitis C virus Real Time Polymerase chain Reaction (HCV RT-PCR) — measure level of serum micro ribonucleic acid -122 and insulin resistance in chronic hepatitis C patients using real time polymerase chain reaction
Diagnostic Test: A)fasting serum glucose, B)Fasting serum insulin — measure level of insulin resistance
  Other Names: HOMA-IR scale

SUMMARY:
The hepatitis C virus is a major cause of chronic liver diseases, including cirrhosis and hepatocellular carcinoma, and infects approximately 3 % of the world population (150-170 million). It is estimated that approximately 80 % of patients with acute hepatitis C fail to eliminate the virus and become chronically infected Hepatitis C virus infection is strongly associated with the dysregulation of glucose homoeostasis such as insulin resistance and type 2 diabetes. Despite these findings of insulin resistance development via direct effects on insulin signalling pathway, the complex relationship between intrahepatic Hepatitis C virus infection and extrahepatic insulin resistance remains elusive.

One of the countries most affected by Hepatitis C virus is Egypt. The Egyptian Demographic and Health Surveys measured antibody prevalence among the adult population aged 15-59 years at 10.0% in 2015-substantially higher than global levels.

Several micro ribonucleic acids have been determined to play a key role in regulating viral replication and pathogenesis during infection. micro ribonucleic acid-122 expression is enriched in the liver, accounting for approximately 70 % of the total micro ribonucleic acid population in normal adult hepatocytes. Moreover, a particularly intriguing function of micro ribonucleic acid-122 involves its role in the Hepatitis C virus replication cycle.

Antagonism of micro ribonucleic acid-122 not only reduces viral replication but also reduces Hepatitis C virus propagation by decreasing the expression of enzymes involved in lipid metabolism, which can enhance Hepatitis C virus replication in cell culture models.

DETAILED DESCRIPTION:
The hepatitis C virus (HCV) is an enveloped, single-stranded positive-sense Ribo-Nucleic Acid virus which is a major cause of chronic liver diseases, including cirrhosis and hepatocellular carcinoma (HCC), and infects approximately 3 % of the world population(150-170 million).

One of the countries most affected by HCV is Egypt. The Egyptian Demographic and Health Surveys measured antibody prevalence among the adult population aged 15-59 years at 14.7% in 2009 and at 10.0% in 2015 To attend to this challenge, Egypt developed a national strategy for Hepatitis C Virus control and established HCV prevention and treatment programs using Direct Acting-Antivirals (DAAs).

Egypt launched an ambitious national HCV treatment program aiming to treat over 250,000 chronically infected individuals per year, with the goal of achieving a national chronic infection prevalence of <2% by 2025.

Although the consequences of chronic HCV infection are generally associated with liver manifestations such as hepatic fibrosis, cirrhosis, steatosis (known as non-alcoholic fatty liver disease, NAFLD) and HCC, the liver-related mortality of 350,000 individuals annually is still underestimated due to the lack of consideration of extrahepatic effect including a growing evidence showing that HCV infection is strongly associated with the dysregulation of glucose homoeostasis such as insulin resistance (IR) and type 2 diabetes (T2D).

HCV-related type 2 diabetes mellitus may arise from a complex interaction between IR, steatosis and inflammatory processes People infected with HCV are 4 times more likely to develop Type 2 Diabetes; and HCV-infected patients with uncontrolled glucose are at higher risk to develop advanced liver fibrosis, HCC, and exhibit decreased sustained virologic response (SVR) to traditional interferon treatment.

HCV protein NS5A and the core protein directly inhibit microsomal triglyceride transfer protein (MTP) activity, thereby reducing very low-density lipoprotein (VLDL) assembly and inducing hepatic steatosis.

Over time, accumulation of hepatic triglycerides leads to hepatic IR via decreased insulin-stimulated glycogen synthesis and enhanced hepatic gluconeogenesis; such conditions further cause peripheral IR in multiple organs through increased circulating insulin and free fatty acid levels.

Regarding the molecular mechanisms of regulation of insulin signaling by HCV infection. HCV core protein has been found to increase serine rather than tyrosine phosphorylation of IRS-1 ( insulin Receptor Substrate-1) in hepatocytes, resulting in its degradation and impaired downstream signaling Protien Kinase B signalling pathway.

HCV core protein also stimulates Insulin Receptor Substrate-1 serine phosphorylation via increasing mTOR (mammalian Target Of Rapamycin)levels, resulting in decreased Protien Kinase B signaling.

Reduced surface expression of glucose transporters GLUT1 and GLUT2 with consequential reduction in glucose uptake in HCV-infected hepatocytes has also been reported.

Despite these findings of IR development via direct effects on insulin signaling pathways, the complex relationship between intrahepatic HCV infection and extrahepatic IR remains elusive.

Several miRNAs have been determined to play a key role in regulating viral replication and pathogenesis during HCV infection.

Host miRNAs can be activated by viral integration in the host genome; viral miRNAs can target host mRNAs, , or host miRNAs can target viral mRNAs.

miR-122 expression is enriched in the liver, accounting for approximately 70 % of the total miRNA population in normal adult hepatocytes with approximately 66,000 copies per cell.

miR-122 has a role in the HCV replication cycle, where it binds to two target sites (S1 and S2) in the highly conserved 5' untranslated region of the HCV genome, thus forming a complex of HCV oligomeric miR-122 that protects the HCV genome from nucleolytic degradation as well as from the host innate immune response.

Many metabolic processes are potentially targeted by miR-122, including protein metabolism, carbohydrate metabolism, lipid metabolism and phospholipid metabolism. Signaling pathway ontology revealed several IR-related pathways [eg insulin/Insulin Growth Factor/Protien Kinase B signaling, Phosphoinositide 3-Kinase signaling, apoptosis, Epidermal Growth Factor receptor signaling,G protien-coupled receptors signaling pathway.

Antagonism of miRNA-122 not only reduces viral replication but also reduces HCV propagation by decreasing the expression of enzymes involved in lipid metabolism, which can enhance HCV replication in cell culture models.

miR-122 represents an interesting therapeutic target for the treatment of liver disease including viral hepatitis, fibrosis, steatosis and HCC. Experimental studies have elegantly demonstrated that a miR-122 inhibitor efficiently reduces viral load in chronically infected HCV patients without detectable resistance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV patients eligible for treatment with Direct Acting Antivirals.
* Chronic HCV patients 3 months after starting of treatment

Exclusion Criteria:

* Cirrhosis
* Diabetes Mellitus
* Hemochromatosis
* HBV
* HIV
* Hepatocellular carcinoma (HCC)
* Chemotherapy
* Organ transplantation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on chronic HCV patients attending the out patient AlRajhy Liver Institute Sovaldi Clinic who are not known to be diabetics
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of change in the level of serum micro ribonucleic acid-122 in Chronic Hepatitis C patients | 3 months
  Measure the level of micro ribonucleic acid-122 on the viral load of chronic hepatitis C patients treated with Sofosbuvir/Daclatasvir regimen using Real Time Polymerase Chain Reaction

CONTACTS AND LOCATIONS:
Overall Officials: Riham A Abdelmegid, MD, Principal Investigator — Assiut University, Faculty of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singhal A, Agrawal A, Ling J. Regulation of insulin resistance and type II diabetes by hepatitis C virus infection: A driver function of circulating miRNAs. J Cell Mol Med. 2018 Apr;22(4):2071-2085. doi: 10.1111/jcmm.13553. Epub 2018 Feb 7. PMID 29411512
- [Background] Kouyoumjian SP, Chemaitelly H, Abu-Raddad LJ. Characterizing hepatitis C virus epidemiology in Egypt: systematic reviews, meta-analyses, and meta-regressions. Sci Rep. 2018 Jan 26;8(1):1661. doi: 10.1038/s41598-017-17936-4. PMID 29374178